CLINICAL TRIAL: NCT04956861
Title: HIV-1, Insufficient Sleep and Vascular Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Christopher DeSouza, Professor, University of Colorado, Boulder
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 150465
Record Dates: First submitted 2021-06-23; First posted 2021-07-09 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: HIV-1
Keywords: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (No Intervention): Phase 1 is a cross-sectional study to compare endothelial vasodilator and fibrinolytic function in ART-treated HIV-1-seropositive adults who habitually sleep more than 7 hours/night (normal sleep) and those who habitually sleep less than 7 hours/night (short sleep).
- Phase 2 (Experimental): Phase 2 is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator and fibrinolytic function in ART-treated HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
  Interventions: Behavioral: Individualized Targeted Sleep

INTERVENTIONS:
Behavioral: Individualized Targeted Sleep — The investigators will employ an 8-week individualized targeted sleep intervention. Individualized targeted interventions have the advantage of improving adherence, reducing attrition, and making the strategy personally meaningful.
  Arms: Phase 2

SUMMARY:
The investigators hypothesize that chronic insufficient sleep is associated with diminished endothelium-dependent nitric oxide-mediated vasodilation and tissue-type plasminogen activator release in anti-retroviral (ART)-treated HIV-1-seropositive adults. Furthermore, the investigators hypothesize that the postulated diminishment in endothelial vasodilator and fibrinolytic function with insufficient sleep will be due, at least in part, to increased oxidative stress. Moreover, increasing sleep duration and improving sleep quality will increase both endothelium-dependent nitric oxide-mediated vasodilation and endothelial tissue-type plasminogen activator release in ART-treated HIV-1-seropositive adults. Increases in endothelial vasodilator and fibrinolytic function will be due, at least in part, to reduced oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women of all races and ethnic backgrounds aged 40-75 years with documented HIV-1 infection.
* Subjects will be HIV-1-seropositive individuals on a stable DHHS approved ART regimen for at least 6 months, with documented virologic suppression (<50 copies HIV-1 RNA/mL) for at least 3 months.
* All subjects must have CD4+ T cell counts >200 cells/mm3 at the time of study entry.
* Subjects will be free of overt CVD as assessed by: a) medical history; b) physical examination; c) electrocardiogram and BP at rest and maximal exercise; d) complete blood chemistries, lipid and lipoprotein, glucose, insulin and hematological evaluation.
* All candidates will be sedentary as determined from the Stanford Physical Activity Questionnaire (<35 kcal/wk) and will not have engaged in any program of regular physical activity for at least 6 months prior to the study.

Exclusion Criteria:

* Receiving hormone replacement therapy (HRT) currently or in the preceding 3-year period.
* Pre- or peri-menopausal women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher DeSouza, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- UC-Boulder Clinical and Translational Research Center, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on the participants nightly sleep duration they were enrolled either in Phase 1: No Intervention: Normal Sleep Group or Phase 1: No Intervention: Short Sleep Group. 10 participants with short nightly sleep duration were recruited separately and enrolled into Phase 2. After participants sign the informed consent, they complete a blood draw and a graded exercise stress test.
Groups:
- No Intervention: Phase 1 Normal Sleep Group; No Intervention: Phase 1 Short Sleep Group: Phase 1 is a cross-sectional study designed to compare endothelial vasodilator (forearm blood flow) and fibrinolytic function (t-PA release) in ART-treated HIV-1-seropositive adults who habitually sleep more than 7 hours/night (normal sleep) and those who habitually sleep less than 7 hours/night (short sleep).
- Experimental: Phase 2: Phase 2 is an intervention study designed to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator (forearm blood flow) and fibrinolytic function (t-PA release) in ART-treated HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
  .
Period: Overall Study
Arm/Group | No Intervention: Phase 1 Normal Sleep Group | No Intervention: Phase 1 Short Sleep Group | Experimental: Phase 2
Started | 36 | 42 | 10
Completed | 28 | 33 | 7
Not Completed | 8 | 9 | 3
Not completed — Withdrawal by Subject | 4 | 4 | 2
Not completed — Physician Decision | 4 | 5 | 1

BASELINE CHARACTERISTICS:
Population: After participants sign the informed consent, they complete a blood draw and a graded exercise stress test. Based on the participants nightly sleep duration they were either in Phase 1: No Intervention: Normal Sleep Group or Phase 1: No Intervention: Short Sleep Group. 10 participants with short nightly sleep duration were recruited separately and enrolled in Phase 2. These 10 participants are only counted in the Phase 2 Sleep Intervention Study.
Groups:
- Experimental: Phase 2 Sleep Intervention Study: Phase 2 is an intervention study designed to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator (forearm blood flow) and fibrinolytic function (t-PA release) in ART-treated HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
- Total: Total of all reporting groups
Arm/Group | No Intervention: Phase 1 Normal Sleep Group | No Intervention: Phase 1 Short Sleep Group | Experimental: Phase 2 Sleep Intervention Study | Total
Number analyzed (Participants) | 36 | 42 | 10 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 42 | 10 | 88
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 13
  Male | 31 | 36 | 8 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 4 | 14
  Not Hispanic or Latino | 31 | 37 | 6 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 34 | 39 | 10 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 42 | 10 | 88

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Forearm Blood Flow (FBF) Response to Acetylcholine (ACh)
Description: FBF was measured via strain-gauge venous occlusion plethysmography in response to saline for 5 minutes and then to ACh (4.0, 8.0 and 16.0 ug/100 mL tissue/min; the doses of Acetylcholine infused into the brachial artery) for 5 minutes at each dose. Flows during the last minute of saline and each drug dose were measured and the mean value reported.
  Values after saline and after ACh 4.0, 8.0 and 16.0 at week 3 are reported.
Time Frame: FBF response to ACh will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Population: The number or participants analyzed is different than the participant flow module as these are the participants who completed visit 3.
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Normal Sleep Duration: Normal Sleep Duration group slept >7 h/night.
- Short Sleep Duration: Short Sleep Duration group slept <7h/night.
Arm/Group | Normal Sleep Duration | Short Sleep Duration
Number analyzed (Participants) | 18 | 22
mL/100 mL tissue/min
  Saline | 4.6 (0.3) | 4.2 (0.3)
  ACh 4.0 | 11.7 (0.8) | 9.9 (0.5)
  ACh 8.0 | 12.4 (0.8) | 10.5 (0.6)
  ACh 16.0 | 14.1 (0.7) | 12.0 (0.6)

2. Primary Outcome: Phase 2: FBF Response to Acetylcholine (ACh)
Description: FBF to ACh will be measured following the participants 8 week sleep intervention.
Time Frame: FBF response to ACh will be measured during Phase 2 at the participants visit 9 which is ~11 weeks from their respective start date
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Phase 2 Before Sleep Intervention: Phase 2 is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator and fibrinolytic function in Anti-retroviral-treated (ART) HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
- Phase 2 After Sleep Intervention: Phase 2 is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator and fibrinolytic function in Anti-retroviral-treated (ART) HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
  Individualized Targeted Sleep: The investigators will employ an 8-week individualized targeted sleep intervention. Individualized targeted interventions have the advantage of improving adherence, reducing attrition, and making the strategy personally meaningful.
Arm/Group | Phase 2 Before Sleep Intervention | Phase 2 After Sleep Intervention
Number analyzed (Participants) | 7 | 7
mL/100 mL tissue/min
  Saline | 4.2 (0.4) | 4.0 (0.3)
  ACh 4.0 | 9.2 (0.8) | 11.1 (0.7)
  Ach 8.0 | 9.9 (0.9) | 12.2 (0.7)
  Ach 16.0 | 11.3 (0.9) | 14.0 (0.6)

3. Primary Outcome: Phase 1: Forearm Blood Flow (FBF) Response to Sodium Nitroprusside (NTP)
Time Frame: FBF response to NTP will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Population: The number or participants analyzed is different than the participant flow module due to availability of Sodium Nitroprusside.
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Arm/Group | Normal Sleep Duration | Short Sleep Duration
Number analyzed (Participants) | 18 | 22
mL/100 mL tissue/min
  Saline | 4.8 (0.4) | 4.0 (0.3)
  NTP 1.0 | 13.9 (0.9) | 12.4 (0.8)
  NTP 2.0 | 16.1 (1.0) | 14.5 (0.7)
  NTP 4.0 | 17.0 (1.1) | 16.7 (0.8)

4. Primary Outcome: Phase 2: Forearm Blood Flow (FBF) Response to Sodium Nitroprusside (NTP)
Description: FBF to NTP will me measured following the participants 8 week sleep intervention
Time Frame: FBF response to NTP will be measured during Phase 2 at the participants visit 9 which is ~11 weeks from their respective start date
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Phase 2 Before Sleep Intervention: Phase 2 is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator and fibrinolytic function in ART-treated HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
- Phase 2 After Sleep Intervention: Phase 2 is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator and fibrinolytic function in ART-treated HIV-1-seropositive adults who habitually sleep less than 7 hours/night.
  Individualized Targeted Sleep: The investigators will employ an 8-week individualized targeted sleep intervention. Individualized targeted interventions have the advantage of improving adherence, reducing attrition, and making the strategy personally meaningful.
Arm/Group | Phase 2 Before Sleep Intervention | Phase 2 After Sleep Intervention
Number analyzed (Participants) | 7 | 7
mL/100 mL tissue/min
  Saline | 3.6 (0.4) | 4.2 (0.6)
  NTP 1.0 | 12.0 (0.9) | 13.8 (1.1)
  NTP 2.0 | 13.9 (0.9) | 14.6 (1.2)
  NTP 4.0 | 15.7 (1.1) | 15.7 (1.4)

5. Primary Outcome: Phase 1: Endothelial Tissue Type Plasminogen Activator (t-PA) Release in Response to Bradykinin (BDK)
Description: Net endothelial release of t-PA antigen in response to BDK was calculated using the following equation:
  Net release = (Cv-Ca) x (FBF x [101-hematocrit/100]) where Cv and Ca represent the concentration in the vein and artery respectively. A positive difference indicated a net release and a negative difference, net uptake. Arterial and venous blood samples were collected simultaneously at the end of saline and each dose of BDK (12.5, 25.0 and 50.0 ng/100mL tissue/min). Enzyme immunoassay was used to determine t-PA antigen concentrations. Hematocrit was measured in triplicate using the standard microhematocrit technique and corrected for trapped plasma volume within the red blood cells.
Time Frame: t-PA release will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Population: The number of participants analyzed is different than reported in the participant flow module due to the availability of BDK during the clinical trial.
Measure: Mean (Standard Error); unit: ng/100 mL tissue/min
Arm/Group | Normal Sleep Duration | Short Sleep Duration
Number analyzed (Participants) | 16 | 14
ng/100 mL tissue/min
  Saline | -0.8 (0.6) | -1.0 (0.5)
  BDK 12.5 | 20.9 (3.2) | 11.4 (2.8)
  BDK 25.0 | 33.3 (4.7) | 23.8 (3.2)
  BDK 50.0 | 53.5 (7.6) | 33.4 (4.1)

6. Primary Outcome: Phase 2: Endothelial t-PA Release in Response to Bradykinin (BDK)
Description: Endothelial t-PA release will me measured following the participants 8 week sleep intervention. Net endothelial release of t-PA antigen in response to BDK was calculated using the following equation:
  Net release = (Cv-Ca) x (FBF x [101-hematocrit/100]) where Cv and Ca represent the concentration in the vein and artery respectively. A positive difference indicated a net release and a negative difference, net uptake. Arterial and venous blood samples were collected simultaneously at the end of saline and each dose of BDK (12.5, 25.0 and 50.0 ng/100mL tissue/min). Enzyme immunoassay was used to determine t-PA antigen concentrations. Hematocrit was measured in triplicate using the standard microhematocrit technique and corrected for trapped plasma volume within the red blood cells.
Time Frame: t-PA release will be measured during Phase 2 at the participants visit 9 which is ~11 weeks from their respective start date
Measure: Mean (Standard Error); unit: ng/100 mL tissue/min
Arm/Group | Phase 2 Before Sleep Intervention | Phase 2 After Sleep Intervention
Number analyzed (Participants) | 5 | 5
ng/100 mL tissue/min
  Saline | -1.8 (1.8) | -2.1 (2.5)
  BDK 12.5 | 15.1 (7.1) | 25.4 (5.8)
  BDK 25.0 | 20.6 (6.3) | 50.1 (14.6)
  BDK 50.0 | 38.9 (8.4) | 78.8 (16.6)

7. Primary Outcome: Phase 1: FBF Response to ACh+Ng-monomethyl-L-arginine (L-NMMA)
Description: To determine the contribution of nitric oxide to ACh-mediated vasodilation, FBF to ACh was quantified before and after infusion of L-NMMA. After ACh was infused as described in Outcome measure 1 the ACh dose response was repeated with the continuous infusion of L-NMMA.
Time Frame: FBF response to ACh+L-NMMA will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Normal Sleep Duration (ACh): Normal Sleep Duration group slept >7 h/night.
  Forearm blood flow (FBF) measured in response to Acetylcholine.
- Normal Sleep Duration (ACh+L-NMMA): Normal Sleep Duration group slept >7 h/night.
  FBF measured in response to Acetylcholine+L-NMMA.
- Short Sleep Duration (ACh): Short Sleep Duration group slept <7h/night.
  Forearm blood flow (FBF) measured in response to Acetylcholine.
- Short Sleep Duration (ACh+L-NMMA): Short Sleep Duration group slept <7h/night.
  FBF measured in response to Acetylcholine+L-NMMA.
Arm/Group | Normal Sleep Duration (ACh) | Normal Sleep Duration (ACh+L-NMMA) | Short Sleep Duration (ACh) | Short Sleep Duration (ACh+L-NMMA)
Number analyzed (Participants) | 18 | 18 | 22 | 22
mL/100 mL tissue/min
  Saline | 4.6 (0.3) | 4.0 (0.3) | 4.2 (0.3) | 3.3 (0.2)
  ACh 4.0 | 11.7 (0.8) | 9.2 (0.8) | 9.9 (0.5) | 8.8 (0.5)
  ACh 8.0 | 12.4 (0.8) | 9.9 (0.8) | 10.6 (0.6) | 9.6 (0.6)
  ACh 16.0 | 14.1 (0.7) | 12.1 (0.8) | 12.0 (0.6) | 11.1 (0.6)

8. Primary Outcome: Phase 1: FBF Response to ACh+Vitamin C
Description: After allowing sufficient time (45 minutes) for FBF to return to levels similar to that of saline Vitamin C was infused at a constant rate (12 mg/100 mL tissue/min) for 5 minutes. This vitamin C concentration has been show to improve endothelium dependent vasodilation in conditions associated with oxidative stress. Vitamin C infusion was maintained at the same rate while the ACh dose response was repeated.
Time Frame: FBF response to ACh+Vitamin C will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Normal Sleep Duration (ACh+Vitamin C): Normal Sleep Duration group slept >7 h/night.
  FBF measured in response to Acetylcholine+Vitamin C.
- Short Sleep Duration (ACh+Vitamin C): Short Sleep Duration group slept <7h/night.
  FBF measured in response to Acetylcholine+Vitamin C.
Arm/Group | Normal Sleep Duration (ACh) | Normal Sleep Duration (ACh+Vitamin C) | Short Sleep Duration (ACh) | Short Sleep Duration (ACh+Vitamin C)
Number analyzed (Participants) | 18 | 18 | 22 | 22
mL/100 mL tissue/min
  Saline | 4.6 (0.3) | 5.1 (0.4) | 4.2 (0.3) | 4.4 (0.3)
  Ach 4.0 | 11.7 (0.8) | 14.3 (0.9) | 9.9 (0.5) | 13.3 (0.6)
  Ach 8.0 | 12.4 (0.8) | 15.2 (0.8) | 10.5 (0.6) | 14.0 (0.7)
  Ach 16.0 | 14.1 (0.7) | 16.7 (0.8) | 12.0 (0.6) | 15.9 (0.7)

9. Primary Outcome: Phase 2: FBF Response to ACh+L-NMMA
Description: FBF to ACh+L-NMMA will me measured following the participants 8 week sleep intervention. To determine the contribution of nitric oxide to ACh-mediated vasodilation, FBF to ACh was quantified before and after infusion of L-NMMA. After ACh was infused as described in Outcome measure 1 the ACh dose response was repeated with the continuous infusion of L-NMMA.
Time Frame: FBF response to ACh+L-NMMA will be measured during Phase 2 at the participants visit 9 which is ~11 weeks from their respective start date
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Short Sleep Duration (ACh) Before Intervention: Short Sleep Duration group slept <7h/night.
  Before Intervention: Forearm blood flow (FBF) measured in response to Acetylcholine.
- Short Sleep Duration (ACh+L-NMMA) Before Intervention: Short Sleep Duration group slept <7h/night.
  Before Intervention: FBF measured in response to Acetylcholine+L-NMMA.
- Short Sleep Duration (ACh) After Intervention: Short Sleep Duration group slept <7h/night.
  After Intervention: Forearm blood flow (FBF) measured in response to Acetylcholine.
- Short Sleep Duration (ACh+L-NMMA) After Intervention: Short Sleep Duration group slept <7h/night.
  After Intervention: FBF measured in response to Acetylcholine+L-NMMA.
Arm/Group | Short Sleep Duration (ACh) Before Intervention | Short Sleep Duration (ACh+L-NMMA) Before Intervention | Short Sleep Duration (ACh) After Intervention | Short Sleep Duration (ACh+L-NMMA) After Intervention
Number analyzed (Participants) | 7 | 7 | 7 | 7
mL/100 mL tissue/min
  Saline | 4.2 (0.4) | 3.3 (0.3) | 4.0 (0.3) | 3.8 (0.5)
  ACh 4.0 | 9.2 (0.8) | 9.0 (0.8) | 11.1 (0.7) | 7.6 (0.6)
  ACh 8.0 | 9.9 (0.9) | 9.7 (0.9) | 12.2 (0.7) | 10.1 (1.1)
  ACh 16.0 | 11.3 (0.9) | 10.8 (0.9) | 14.0 (0.6) | 10.8 (1.0)

10. Primary Outcome: Phase 2: FBF Response to ACh+Vitamin C
Description: FBF to ACh+Vitamin C will me measured following the participants 8 week sleep intervention. After allowing sufficient time (45 minutes) for FBF to return to levels similar to that of saline Vitamin C was infused at a constant rate (12 mg/100 mL tissue/min) for 5 minutes. This vitamin C concentration has been show to improve endothelium dependent vasodilation in conditions associated with oxidative stress. Vitamin C infusion was maintained at the same rate while the ACh dose response was repeated.
Time Frame: FBF response to ACh+Vitamin C will be measured during Phase 2 at the participants visit 9 which is ~11 weeks from their respective start date
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Groups:
- Short Sleep Duration (ACh+Vitamin C) Before Intervention: Short Sleep Duration group slept <7h/night.
  Before Intervention: FBF measured in response to Acetylcholine+Vitamin C.
- Short Sleep Duration (ACh+Vitamin C) After Intervention: Short Sleep Duration group slept <7h/night.
  After Intervention: FBF measured in response to Acetylcholine+Vitamin C.
Arm/Group | Short Sleep Duration (ACh) Before Intervention | Short Sleep Duration (ACh+Vitamin C) Before Intervention | Short Sleep Duration (ACh) After Intervention | Short Sleep Duration (ACh+Vitamin C) After Intervention
Number analyzed (Participants) | 7 | 7 | 7 | 7
mL/100 mL tissue/min
  Saline | 4.2 (0.4) | 4.3 (0.5) | 4.0 (0.3) | 4.8 (0.6)
  ACh 4.0 | 9.2 (0.8) | 12.6 (1.3) | 11.1 (0.7) | 12.4 (1.7)
  ACh 8.0 | 9.9 (0.9) | 13.5 (1.3) | 12.2 (0.7) | 13.0 (1.5)
  ACh 16.0 | 11.3 (0.9) | 14.8 (1.5) | 14.0 (0.6) | 14.2 (1.5)

11. Secondary Outcome: Nightly Sleep Duration
Description: Nightly sleep duration was calculated as the weighted average of weeknights and weekend values [(5 x weekday sleep duration)+(2 x weekend sleep duration)/7].
Time Frame: Baseline
Population: Nightly sleep duration was measured during Phase 1 at the participants initial visit.
Measure: Mean (Standard Error); unit: hours/night
Arm/Group | Normal Sleep Duration | Short Sleep Duration
Number analyzed (Participants) | 30 | 38
hours/night | 7.8 (0.2) | 5.8 (0.2)

ADVERSE EVENTS:
Time Frame: Data was collected for participants while they were enrolled in the study. Each participant was in the study for a maximum of 4 months.
Description: For simplicity in the reporting of the results with regards to the Adverse Event Table, Phase 1 the normal sleep duration group and the short sleep duration group are combined since no adverse events occurred or were reported.
Groups:
- Phase 1: Cross-sectional Study: Phase 1 is a cross-sectional study to compare endothelial vasodilator (forearm blood flow) and fibrinolytic function (t-PA release) in ART-treated HIV-1-seropositive adults who habitually sleep more than 7 hours/night (normal sleep) and those who habitually sleep less than 7 hours/night (short sleep).
- Phase 2: Intervention Study: Phase 2 is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator (forearm blood flow) and fibrinolytic function (t-PA release) in ART-treated HIV-1-seropositive adults who habitually sleep less than 7 hours/night (short sleep).
  Participants from phase 1 were invited to take part in phase 2.
Arm/Group | Phase 1: Cross-sectional Study | Phase 2: Intervention Study
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/10
Other Adverse Events (participants affected / at risk) | 0/78 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04956861/Prot_SAP_000.pdf